CLINICAL TRIAL: NCT04900051
Title: Clinical Efficacy and Safety of Fecal Microbiota Transplantation
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Keimyung University Dongsan Medical Center (Other)
Responsible Party: Principal Investigator, YooJin Lee, Assistant Professor, Keimyung University Dongsan Medical Center
Other Study IDs: 2020-08-016
Record Dates: First submitted 2021-03-31; First posted 2021-05-25 (Actual); Last update posted 2021-05-25 (Actual); Status verified 2021-03

CONDITIONS: Fecal Microbiota Transplantation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Biospecimen Retention: Samples With DNA — Blood laboratory test(CBC, CRP, protein/albumin, AST/ALT, GTP, Total bilirubin/Direct bilirubin), Fecal calprotectin, Stool
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Changes in the fecal microbiota are known to be involved in the etiology of several diseases. The purpose of this study is to evaluate the effectiveness and safety of fecal microbiota transplantation (FMT) in diseases known to be associated with intestinal microbial inbalance. .

DETAILED DESCRIPTION:
This registry will prospectively enroll 300 patients who undergo fecal microbiota transplantation(FMT) at 3 clinical center (Yeungnam university mecial center, Kyungpook national university hospital, Keimyung university dongsan medical center). Feces received from healthy donors are prepared as frozen feces according to a standardized protocol, and transplanted to recipients within 3 months. Next generation sequencing(NGS) is used to check the characteristics of the fecal microbiota of the donor stool, and to evaluate the efficacy by checking the change in the fecal microbium of recipient before and after transplantation. The data is documented for following diseases known to be related to microbium imbalance.

1. Recurrent or Refractory CDI Abdominal symptoms questionnaires, blood laboratory test(CBC, CRP, protein/albumin, AST/ALT, GTP, Total bilirubin/Direct bilirubin)
2. Irritable bowel syndrome, Functional dyspepsia Abdominal symptoms questionnaires, IBS diagnosis and food-related questionnaires, blood laboratory test(CBC, CRP, protein/albumin, AST/ALT, GTP, Total bilirubin/Direct bilirubin)
3. Inflammatory Bowel Disease Abdominal symptoms questionnaires, blood laboratory test(CBC, CRP, protein/albumin, AST/ALT, GTP, Total bilirubin/Direct bilirubin), fecal calprotectin, Colonoscopic examination(Mayo endoscopic subscore, CD-SES)
4. Non-alcoholic steatohepatitis, NASH Abdominal symptoms questionnaires, blood laboratory test(CBC, CRP, protein/albumin, AST/ALT, GTP, Total bilirubin/Direct bilirubin), BMI check
5. Obesity Abdominal symptoms questionnaires, blood laboratory test(CBC, CRP, protein/albumin, AST/ALT, GTP, Total bilirubin/Direct bilirubin), BMI check

ELIGIBILITY:
Inclusion Criteria:

* Those who have been diagnosed with disease to be studied and do not respond to exist treatments

  1. Ulcerative colitis, Crohn disease : Patient who does not responding to anti- TNF treatment for more than 3 month.
  2. Irritable bowel syndrome, Functional dyspepsia : Patient who does not responding to pharmacological therapies and serotonin uptake inhibitor for more than 6 month.
  3. Recurrent of Refractory CDI, NASH, Obesity : Patient who does not responding to treatment for more than 6 month.

Exclusion Criteria:

* Neutrophil (<0.5 x 10*9/L)
* Leukocytosis (> 30.0 x 10*9/L)
* Toxic megacolon confirmed in abdomen Xray
* Pregnant or lactating women

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: * Hospitalized and outpatient aged from 18 to 80 years old
  * Those who agrees after hearing the explanation on the efficacy and safety of fecal microbiota transplantation
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-12-24 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Set up a FMT registry | 3 years
  Set up a registry of FMT in diseases known to be associated with intestinal microbial imbalance

SECONDARY OUTCOMES:
Patient outcome of FMT | 6 month
  Compare the severity of diseases, any adverse event before and after FMT
Developing biobank of FMT | 3 Years
  Collect the study sample of microbium from donors and recipients

CONTACTS AND LOCATIONS:
Overall Officials: Lee Yoo Jin, Professor, Principal Investigator — Keimyung University Dongsan Medical Center
Locations (1):
- KeimyungUniversity, Daegu, Jung-gu, South Korea

IPD SHARING:
Plan to Share IPD: No